CLINICAL TRIAL: NCT05533892
Title: Nocardia Rubra Cell Wall Skeleton Plus Hepatic Arterial Infusion Chemotherapy, Lenvatinib and Tislelizumab for Advanced Hepatocellular Carcinoma: a Single-center, Single-arm, Non-randomized Clinical Study
Brief Title: Nocardia Rubra Cell Wall Skeleton (N-CWS) Plus HAIC, Lenvatinib and Tislelizumab in Treating Patients With Advanced HCC
Acronym: CCGLC-007
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wan-Guang Zhang (Other)
Collaborators: Chinese Cooperative Group of Liver Cancer (Other); Chen Xiao-ping Foundation for the Development of Science and Technology of Hubei Province (Other); M&R Pharm (Unknown); Geneplus-Beijing Co. Ltd. (Industry); Yuce Biotechnology Co., Ltd. (Unknown); Geneis (Unknown); Simcere Pharmaceutical Co., Ltd (Other); BeiGene (Industry); Haplox Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Wan-Guang Zhang, Executive Deputy Director of Hepatic Surgery Center, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-S038
Record Dates: First submitted 2022-09-04; First posted 2022-09-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cell wall skeleton, Nocardia; lenvatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nocardia rubra cell wall skeleton (N-CWS) Plus HAIC, Lenvatinib and Tislelizumab (Experimental): N-CWS 400μg hypodermic injected every week (Q1W) for 4 weeks, following by N-CWS 400μg hypodermic injected Q4W. Hepatic arterial infusion of oxaliplatin , fluorouracil, and leucovorin every 3 weeks. Lenvatinib 12 mg (or 8 mg) once daily (QD) oral dosing. Tislelizumab 200mg intravenously every 3 weeks.
  Interventions: Drug: Nocardia rubra cell wall skeleton; Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Nocardia rubra cell wall skeleton — Nocardia rubra cell wall skeleton (N-CWS) 400μg hypodermic injected every 1 week (Q1W) for 4 weeks, following by N-CWS 400μg hypodermic injected every 4 weeks (Q4W)
  Other Names: N-CWS
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks
  Other Names: HAIC
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing
  Other Names: JieLiEn
Drug: Tislelizumab — 200mg intravenously every 3 weeks
  Other Names: BaiZeAn

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nocardia rubra cell wall skeleton plus hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin, lenvatinib and tislelizumab in patients with advanced hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following criteria

* Subjects volunteer to participate in the study and agree to sign the informed consent with good compliance and follow-up.
* Subjects are 18 years old or older when signing the informed consent and gender is not limited.
* Subjects were diagnosed with advanced hepatobiliary malignant tumors (clinical stage IV) by imaging and histological examination, including hepatocellular carcinoma, cholangiocarcinoma, ampullary carcinoma, gallbladder carcinoma and mixed carcinoma.
* The disease is not suitable for radical surgery and/or topical treatment, or disease progression occurs after surgery and/or local treatment.
* At least one measurable lesion (according to mRECIST): the measurable lesion has a long diameter ≥ 10 mm or lymphadenpathy has a short diameter ≥ 15 mm in spiral CT scan.
* Patients fail after at least one systemic failure, including surgery, intervention, radiotherapy, chemotherapy and targeted therapy and require palliative treatment.
* Definition of treatment failure: Disease progression during treatment or relapse after treatment, such as after at least once radical or palliative resection surgery, revenue recurrence or progression after intervention therapy or radiotherapy. Intervention therapy or oxaliplatin treatment must be more than 1 cycle, and molecular targeted therapy must more than ≥14 days.
* Definition of intolerance: Grade ≥IV hematologic toxicity, or grade ≥III non- hematologic toxicity, or grade ≥ II damage of heart, liver and kidney during treatment.
* The ECOG score is 0-2 within 1 week before enrollment.
* Liver function assessment: Child-Pugh Grade A or mild Grade B (≤ 7 points), BCLC stage B-C.
* More than 2 weeks from first-line system treatment failure to sign informed consent for this study, and adverse events returned to normal (NCI-CTCAE ≤ I).
* Estimated survival time ≥ 6 months.
* HBV DNA <2000 IU/ml (104 copies/ml).
* Hematology and organ function are sufficient based on the following laboratory results within 14 days prior to the treatment of this study:
* Whole blood cell examination (no blood transfusion within 14 days, no G-CSF use and no drugs use): Hb≥90g/L, ANC≥1.5×10*9/L, PLT≥80×10*9/L.
* Biochemical examination (no ALB infused within 14 days): ALB≥29 g/L, ALT and AST<5×ULN, TBIL≤1.5×ULN, creatinine≤1.5×ULN (only one of albumin and bilirubin has 2 points with Child-Pugh score).
* Tumor tissue must be available for biomarker analysis prior to the first dose of treatment, If not available, participants can consult the investigator for enrollment agreement.
* Note: If an unstained section is submitted, the new section should be submitted to the laboratory within 14 days.

Exclusion Criteria: Subjects with one or more than one of the following criteria should be excluded

* Clinical stage I-III, and/or with any of the following:
* Suitable for radical surgery,
* Or, without an assessment lesion after radical surgery,
* Or, never receive any first line treatment,
* Or, liver transplantation history or ready for liver transplantation.
* ECOG score ≥ 3 points.
* Received any topical treatment within 4 weeks prior to the study, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection.
* Ascites with clinical symptoms which requires abdominal puncture or drainage therapy, or Child-Pugh score >2.
* With serious systemic diseases such as heart disease and cerebrovascular disease, and the condition is unstable or uncontrollable.
* Already known active central nervous system metastasis and/or cancerous meningitis. Subjects with stable brain metastases after previous treatment may participate as long as no radiologic evidence of progression lasts for at least four weeks prior to this trial and any neurological symptoms have returned to baseline, and no new or enlarged metastatic evidence in brain and no steroids use for at least 7 days prior to trial treatment. Cancer meningitis should be excluded regardless of clinical stability.
* Surgery was performed within 4 weeks prior to the trial and patients must be
* evaluated after wound healing.
* Hepatic and renal dysfunction evidence: jaundice, ascites, and/or bilirubin ≥ 1.5 × ULN, and/or alkaline phosphatase ≥ 3 × ULN, and/or ≥ 3 grade (CTC-AE 5.0) proteinuria (> 3.5g /24 hours), or renal failure requiring blood dialysis or peritoneal dialysis.
* Urine examination shows urinary protein ≥ ++ or 24 hours urine protein >1.0g. Persistent >2 grade (CTCAE5.0) infection.
* History of allogeneic tissue transplantation or solid organ transplantation.
* History of active tuberculosis, such as mycobacterium tuberculosis.
* Intolerant of any drug (or any excipient) in this trial.
* Female patients who are pregnant, breastfeeding or refuse contraception.
* Known or untreated brain metastases, or patients with epilepsy who need medication treatment.
* Patients with bone metastases received palliative radiotherapy (radiation area > 5% bone marrow area) within 4 weeks prior to this study, or there were wounds, ulcers or fractures that could not be healed, or patients have organ transplantation history.
* Gastrointestinal bleeding history in the past 6 months or tendency to gastrointestinal bleeding, such as esophageal varices, local active ulceration lesions, fecal occult blood ≥ (++) (gastroscopy is required when fecal occult blood is (+)).
* Evidence or history of ≥3 grade (CTCAE5.0) bleeding events.
* History of human immunodeficiency virus infection.
* History of hepatitis B virus or hepatitis C virus infection, and not receive regular treatment.
* Severe non-healing wounds, ulcers or fractures.
* Prior treatment with either lenvatinib or any kind of anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs.
* There were no active autoimmune diseases that require systemic treatment such as disease modifying drugs, corticosteroids or immunosuppressants in the past 2 years. Alternative therapies with thyroxine, insulin or corticosteroid are not considered as systemic therapy.
* Diagnosis of immunodeficiency or systemic steroid therapy or any form of immunosuppressants therapy within 7 days prior to this study. A physiological dose of corticosteroids (no more than 7.5 mg/d prednisone or equivalent) can be approved after clinical evaluation.
* There exists drug abuse, or any medical, psychological or social condition which might affect the study, the compliance or even the safety of patients.
* Variable factors which significantly affect drug use and absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction.
* Any >1 grade (CTC-AE5.0) unresolved toxicity due to previous treatment or operation, except for hair loss, anemia, and hypothyroidism.
* Vaccination of any live virus vaccine within 30 days prior to this study, except for seasonal flu vaccines without live virus.
* Previous and current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia and severe impairment of lung function.
* Received a potent CYP3A4 inhibitor treatment within 7 days prior to the study, or received a potent CYP3A4 inducer within 12 days prior to the study.
* Women with fertility agree to abstinence during the treatment period and at least 6 months after the last dose (avoiding heterosexual intercourse) or using a contraceptive method with an annual contraceptive failure rate <1%.
* If a female patient has menstruation and not reached the postmenopausal state (continuously no menstruation ≥ 12 months and no other causes), and has not undergone sterilization by removing the ovaries and/or uterus), then the patient has fertility.
* Contraceptive methods with a contraceptive failure rate <1% include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices.
* The reliability of sexual desire should be evaluated relative to the duration of the clinical trial and lifestyle of patient. Periodic abstinence (eg. calendar days, ovulation, symptomatic body temperature or post-ovulation methods) and in vitro ejaculation are unacceptable methods of contraception.
* Male patients agree to abstinence (no heterosexual intercourse) or use of contraceptive measures and no sperm donation, as defined below:
* When a female partner has fertility, male patients must abstinence from sex during treatment and at least 6 months after the last dose of treatment, or use condoms and other contraceptive methods with contraceptive failure rate <1%. At the same time, male patients must also agree not to donate sperm.
* When a female partner is pregnant, the male patient must abstinence or using a condom during the treatment period and at least 6 months after the last dose of treatment to prevent the fetus from being affected by the study.
* The reliability of sexual desire should be evaluated relative to the duration of the clinical trial and lifestyle of patient. Periodic abstinence (eg. calendar days, ovulation, symptomatic body temperature or post-ovulation methods) and in vitro ejaculation are unacceptable methods of contraception.
* Patients are unsuitable for participation in this research after comprehensive assessment by the researchers.
* Patients participate in another clinical study at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) at 6 months | 6 months
  ORR, as determined based on tumor response according to mRECIST, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.

SECONDARY OUTCOMES:
Overall survival | 6 months
  OS is the length of time from the date of randomization until death from any cause
Adverse events | 6 months
  Safety will be evaluated according to the NCI CTCAE Version 5.0. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.
Progression free survival rate at 6 months | 6 months
  Progression was defined as progressive disease by independent radiologic review according to mRECIST or death from any cause
Duration of response (DOR) | 6 months
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.

CONTACTS AND LOCATIONS:
Overall Officials: Wan-guang Zhang, M.D., Study Chair — Tongji Hospital
Locations (1):
- Hepatic Surgery Center, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No